CLINICAL TRIAL: NCT02711631
Title: Feasibility and Effectiveness of Remote Virtual Reality-Based Cardiac Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Peter Wood, Research Associate, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MedBIKE
Record Dates: First submitted 2015-04-17; First posted 2016-03-17 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Myocardial Infarction
Keywords: coronary angioplasty; cardiac rehabilitation; coronary artery bypass graft
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control: Standard therapy (No Intervention): Participants in this arm of the study will receive standard therapy.
- MedBIKE (Experimental): Participants in this arm will be using the new MedBIKE system as their method of rehabilitation.
  Interventions: Behavioral: MedBIKE

INTERVENTIONS:
Behavioral: MedBIKE — MedBIKE is an exercise cardiac rehabilitation system that allows participants to perform clinical cardiac rehabilitation at home or at a local center, instead of having to travel to the hospital. It provides a high level of physiological monitoring to allow patient safety to be continually monitored while exercising.
  Arms: MedBIKE

SUMMARY:
Regular exercise in patients who have heart disease is highly beneficial and improves quality of life and survival. Exercise training is considered a core component of cardiac rehabilitation (CR), which is a multicomponent program delivered to patients who have heart disease. However, it is severely underutilized because people simply don't have the time or the resources to travel to a CR centre to attend rehab appointments.

The investigators have developed a novel virtual reality (VR) based CR exercise system (MedBike). This system consists of an exercise bike attached to a VR world; it makes exercise engaging and fun. Furthermore, patients can be monitored during exercise remotely over the internet. The investigators intend to perform a pilot randomized controlled trial in which 10 patients are assigned to the MedBike system and 10 to standard CR. The investigators think that the MedBike system will increase exercise program compliance by providing an enjoyable and engaging exercise experience which can be performed in the comfort of one's own home. The investigators think that this will improve fitness (primary endpoint) in these patients. If the investigators demonstrate that home based exercise is feasible, the investigators plan a larger study to prove that it is something that should be broadly implemented in patients with heart disease.

DETAILED DESCRIPTION:
Background Regular exercise, incorporated as part of a comprehensive cardiac rehabilitation (CR) program, improves morbidity and mortality in cardiac patients, especially those with elevated risk profiles. It was reported in a review that exercise decreased all-cause mortality, cardiac mortality, and non-fatal myocardial infarction by 20 to 25%. Of critical importance, CR non-participants exhibit a 30% lower survival rate than those who participate.

Even though exercise training is considered a core component of cardiac rehabilitation it is severely underutilized. The majority of adult patients do not participate in exercise rehabilitation following cardiac events or cardiac surgery; of those eligible, the completion rates are 15% to 30%. Factors associated with poor compliance include greater distance from the hospital, need for transportation (e.g. and parking fees), lack of self motivation, poor social support, low self-esteem, fear of safety and lack of enjoyment. In order to overcome these barriers, researchers and clinicians have been turning toward eHealth solutions to decentralize the CR process, increase accessibility, and potentially increase the comfort and enjoyment derived from exercise. This approach aligns closely with the American Heart Association's recommendation that Internet-based techniques be used to improve the CR experience for both patients and healthcare providers.

The Advanced Man Machine Interface Laboratory (AMMI), University of Alberta has developed a novel virtual reality (VR) enhanced exercise system (MedBIKE) which provides an engaging and enjoyable exercise experience while allowing CR patients to exercise in the comfort of their own home. The system consists of a mountain bike mounted on a wirelessly controlled resistance machine fed directly into a VR console.

This VR console allows for a heightened exercise experience for the patient by allowing them to cycle through a virtual landscape. While exercising, the patients are monitored remotely in real-time by a CR clinician using wireless biometric sensors (electrocardiogram, blood pressure, and pulse oximetry) and a bidirectional audio-video Internet connection. The investigators believe that by enhancing the exercise experience, eliminating distance and transportation issues, and providing ongoing support from key healthcare providers, patient compliance with the CR exercise program will improve. The MedBIKE has not been tested in a clinical trial.

Objective and Hypothesis:

To perform a randomized pilot feasibility study to assess the:

1. Feasibility of having CR patients perform home-based exercise with MedBIKE
2. Effectiveness of the MedBIKE system to improve fitness (as measured by exercise tolerance testing using the Bruce protocol). Since this is a feasibility trial, it will not be fully powered but the investigators will gain preliminary information for a sample size calculation (for a larger trial)
3. Effectiveness of the MedBIKE system to improve patient compliance to CR.

The investigators hypothesize that home-based CR using the MedBIKE system is feasible and will effectively improve fitness and compliance (more frequent exercise sessions and a greater number of total hours). The latter endpoints may not reach statistical significance but the investigators plan a larger funding application to Canadian Institute for Health Research for a properly powered study based upon sample size calculations provided by this pilot randomized control trial.

Methods Adults (age 18y or older) who have had a recent cardiac event, angioplasty or cardiac surgery (within 2 weeks) and who have been referred for CR at the Jim Pattison Centre for Heart Health (JPCHH) will be enrolled in this pilot randomised controlled trial. Consecutive, consenting subjects will be randomised 1:1 (computer based randomisation through an independent clinical trials centre to ensure allocation concealment independent of the study team) to the MedBike system or standard rehabilitation in the JPCHH.

Subjects:

Twenty participants (10 intervention and 10 control) will be enrolled. To avoid enrolling higher risk subjects that require in-person CR supervision, the investigators will exclude subjects with a history of heart failure, cardiomyopathy, severe valvular disease or rhythm disturbances requiring cardioversion. Patients with defibrillators and those unable to consent, speak English, comprehend study procedures, cycle on a stationary bike, perform a treadmill test, or access the internet from home will be excluded.

Controls (Standard CR) The standard cardiac rehab program is 8 weeks in duration, with patients exercising under supervision once per week in the JPCHH. Each session will consist of 30 minutes of cardiorespiratory exercise at a moderate intensity (60 to 80% of predicted heart rate max or maximum effort achieved during an exercise tolerance test) and a 5-minute warm-up and cool down period. Participants will be encouraged to supplement the JPCHH program with an additional optional 2-3 activity sessions per week to be performed in the home or a commercial exercise facility, in accordance with the standard therapy protocol of the JCPHH. No upper limit of training sessions will be set.

Intervention Subjects in the intervention arm will complete the same exercise prescription assigned to the JPCHH patients (i.e.one session will be scheduled per week for 8 weeks as described above). MedBIKE patients will also be encouraged to use the MedBIKE an additional 2-3x/week (these are optional training sessions). No upper limit of training sessions will be set. Scheduled training sessions will be monitored remotely in real-time by a cardiac rehabilitation clinician from the JPCHH via a bidirectional audio-video feed. Biometric information (electrocardiogram, blood pressure, pulse oximetry) will be collected in real time. Monitoring will occur from a clinic room in the JPCHH. Biometric information from the training sessions will be stored on a secure server located within the Faculty of Medicine and Dentistry, University of Alberta. A secure, encrypted, HIPAA compliant data transmission profile will be utilized for patient data transmission, reception and storage.

Additional Care Other elements of protocolized CR including multidisciplinary care will remain unaltered in both groups. This includes a supervised treadmill test performed upon admission to, and discharge from, the JPCHH using the Bruce protocol.

Endpoints:

1. Fitness: Measured at baseline and 8wk in the JPCHH using the Bruce protocol exercise tolerance test. The total time exercised will be determined. For the primary endpoint, similar to prior studies, the investigators will calculate the proportion of patients achieving an increase in 1 min from baseline to 8 weeks and compare this proportion between groups. A 1 min increase corresponds to a 1 to 1.5 metabolic equivalent increase on the Bruce protocol; this translates to a projected 12% to 50% reduction in mortality.
2. Compliance: by comparing the number of scheduled supervised sessions attended (either in the JPCHH [controls] or remotely supervised [intervention]), the self-reported total number exercise sessions participated in, and the cumulative number of hours exercised by each subject. These latter two endpoints will thus include information collected from optional exercise sessions.
3. Change in cardiovascular risk factors from baseline to 8wk: blood pressure (BP), A1c, smoking status, lipids.

Data Collection and Analysis:

Baseline data collection will include age, sex, smoking status, past medical history including cardiovascular risk factors and disease, height, weight, waist circumference, BP, A1c, fasting lipid profile, resting heart rate, and Bruce protocol treadmill time. Follow-up data collection (at 8 weeks) will include updated medical events, weight, waist circumference, BP, A1c, fasting lipids, resting heart rate, follow-up treadmill time, self-reported total number of exercise sessions and hours exercised. Continuous variables will be summarized as means ± standard deviations (SD) and dichotomous variables as counts and proportions. Continuous outcomes will be compared between study arms using logistic regression adjusting for age, sex and unbalanced baseline characteristics (including for the primary endpoint). Linear regression will be used for dichotomous outcomes and Poisson regression for counts.

Sample Size:

The sample size is low, but this is a feasibility trial. Only one CR session per week will be supervised; optional CR sessions will be ascertained through self-report, which is prone to bias. However, to mitigate this, fitness will be assessed through an objective treadmill test.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of stable ischemic heart disease
* received a recent uncomplicated coronary angioplasty or coronary artery bypass graft
* participants will be required to have a referral for cardiac rehabilitation.

Exclusion Criteria:

* a history of heart failure
* a history of cardiac arrhythmia requiring cardioversion
* an implantable cardiac defibrillator
* unable to cycle on a bike

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Fitness | 8 weeks
  Change in fitness measured at 8 weeks using Bruce protocol treadmill test performance time as a metric.
Compliance | 8 weeks
  The investigators will be counting the number of sessions performed in both study arms in their 8 weeks of rehab to determine if there is a difference. This will include scheduled and unscheduled sessions through session documentation and patient self-reporting.

SECONDARY OUTCOMES:
Change in resting blood pressure | 8 weeks
  Change in resting blood pressure (mmHg) will be measured after 8 weeks of cardiac rehab exercise therapy using a 5 BP measurement protocol where 5 BP's (BPtru device) will be taken and the mean will be used.
Change in A1c | 8 weeks
  A change in A1c will be measured at 8 weeks against baseline using a second set of blood taken in the week following the final exercise session.
Smoking status | 8 weeks
  A change in smoking status will be assessed using an interview format following the final cardiac rehab session.
Cholesterol (LDL, HDL, Triglycerides) | 8 weeks
  A change in total and relative cholesterol will be assessed at the end of the 8 weeks of cardiac rehab via a blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Raj S Padwal, MD MSc, Principal Investigator — Division of General Internal Medicine, Faculty of Medicine and Dentistry, University of Alberta; Paolo Raggi, MD, Principal Investigator — Mazankowski Alberta Heart Institute, University of Alberta Hospital
Locations (1):
- Jim Pattison Centre for Heart Health, Mazankowski Heart Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Thompson PD, Buchner D, Pina IL, Balady GJ, Williams MA, Marcus BH, Berra K, Blair SN, Costa F, Franklin B, Fletcher GF, Gordon NF, Pate RR, Rodriguez BL, Yancey AK, Wenger NK; American Heart Association Council on Clinical Cardiology Subcommittee on Exercise, Rehabilitation, and Prevention; American Heart Association Council on Nutrition, Physical Activity, and Metabolism Subcommittee on Physical Activity. Exercise and physical activity in the prevention and treatment of atherosclerotic cardiovascular disease: a statement from the Council on Clinical Cardiology (Subcommittee on Exercise, Rehabilitation, and Prevention) and the Council on Nutrition, Physical Activity, and Metabolism (Subcommittee on Physical Activity). Circulation. 2003 Jun 24;107(24):3109-16. doi: 10.1161/01.CIR.0000075572.40158.77. No abstract available. PMID 12821592
- [Background] Oldridge NB, Guyatt GH, Fischer ME, Rimm AA. Cardiac rehabilitation after myocardial infarction. Combined experience of randomized clinical trials. JAMA. 1988 Aug 19;260(7):945-50. PMID 3398199
- [Background] Jelinek MV, Thompson DR, Ski C, Bunker S, Vale MJ. 40 years of cardiac rehabilitation and secondary prevention in post-cardiac ischaemic patients. Are we still in the wilderness? Int J Cardiol. 2015 Jan 20;179:153-9. doi: 10.1016/j.ijcard.2014.10.154. Epub 2014 Oct 29. PMID 25464436
- [Background] Suaya JA, Shepard DS, Normand SL, Ades PA, Prottas J, Stason WB. Use of cardiac rehabilitation by Medicare beneficiaries after myocardial infarction or coronary bypass surgery. Circulation. 2007 Oct 9;116(15):1653-62. doi: 10.1161/CIRCULATIONAHA.107.701466. Epub 2007 Sep 24. PMID 17893274
- [Background] Bjarnason-Wehrens B, McGee H, Zwisler AD, Piepoli MF, Benzer W, Schmid JP, Dendale P, Pogosova NG, Zdrenghea D, Niebauer J, Mendes M; Cardiac Rehabilitation Section European Association of Cardiovascular Prevention and Rehabilitation. Cardiac rehabilitation in Europe: results from the European Cardiac Rehabilitation Inventory Survey. Eur J Cardiovasc Prev Rehabil. 2010 Aug;17(4):410-8. doi: 10.1097/HJR.0b013e328334f42d. PMID 20300001
- [Background] Neubeck L, Freedman SB, Clark AM, Briffa T, Bauman A, Redfern J. Participating in cardiac rehabilitation: a systematic review and meta-synthesis of qualitative data. Eur J Prev Cardiol. 2012 Jun;19(3):494-503. doi: 10.1177/1741826711409326. PMID 22779092
- [Background] Slovinec D'Angelo ME, Pelletier LG, Reid RD, Huta V. The roles of self-efficacy and motivation in the prediction of short- and long-term adherence to exercise among patients with coronary heart disease. Health Psychol. 2014 Nov;33(11):1344-53. doi: 10.1037/hea0000094. Epub 2014 Aug 18. PMID 25133848
- [Background] Evenson KR, Fleury J. Barriers to outpatient cardiac rehabilitation participation and adherence. J Cardiopulm Rehabil. 2000 Jul-Aug;20(4):241-6. doi: 10.1097/00008483-200007000-00005. PMID 10955265
- [Background] Balady GJ, Ades PA, Bittner VA, Franklin BA, Gordon NF, Thomas RJ, Tomaselli GF, Yancy CW; American Heart Association Science Advisory and Coordinating Committee. Referral, enrollment, and delivery of cardiac rehabilitation/secondary prevention programs at clinical centers and beyond: a presidential advisory from the American Heart Association. Circulation. 2011 Dec 20;124(25):2951-60. doi: 10.1161/CIR.0b013e31823b21e2. Epub 2011 Nov 14. No abstract available. PMID 22082676
- [Background] Pollock ML, Bohannon RL, Cooper KH, Ayres JJ, Ward A, White SR, Linnerud AC. A comparative analysis of four protocols for maximal treadmill stress testing. Am Heart J. 1976 Jul;92(1):39-46. doi: 10.1016/s0002-8703(76)80401-2. PMID 961576
- [Background] Lear SA, Singer J, Banner-Lukaris D, Horvat D, Park JE, Bates J, Ignaszewski A. Randomized trial of a virtual cardiac rehabilitation program delivered at a distance via the Internet. Circ Cardiovasc Qual Outcomes. 2014 Nov;7(6):952-9. doi: 10.1161/CIRCOUTCOMES.114.001230. Epub 2014 Sep 30. No abstract available. PMID 25271050
- [Background] Keteyian SJ, Brawner CA, Savage PD, Ehrman JK, Schairer J, Divine G, Aldred H, Ophaug K, Ades PA. Peak aerobic capacity predicts prognosis in patients with coronary heart disease. Am Heart J. 2008 Aug;156(2):292-300. doi: 10.1016/j.ahj.2008.03.017. Epub 2008 May 22. PMID 18657659